CLINICAL TRIAL: NCT07098182
Title: Clinical Study Evaluating the Contribution of Preserving the Superior Left Colic Artery to the Vascularization of the Descending Colon Prior to Colorectal Anastomosis During Left-Sided or Rectal Resections for Colorectal or Ovarian Cancer. (Revascularisation Colique)
Brief Title: Contribution of Preserving the Superior Left Colic Artery to the Vascularization of the Descending Colon Prior to Colorectal Anastomosis During Left-Sided or Rectal Resections for Colorectal or Ovarian Cancer. (Revascularisation Colique)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2025-03 REV; 2025-A01566-43 (Other: ID-RCB)
Record Dates: First submitted 2025-07-11; First posted 2025-08-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Rectal Cancer; Colon Cancer; Ovarian Cancer
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms; Ovarian Neoplasms | interventions — Constriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): During surgery, on the same patient who received left or colorectal resection with ligation of the lower mesenteric artery below of the emergence of the left colic artery, the steps will be as follows:
  * Time 1: Clamping of the inferior mesenteric artery at its origin (resulting in clamping the left colic artery),
    1. Evaluation of the fluorescence intensity at the area of interest after Indocyanine green injection :
    2. Measurement of the blood pressure of the marginal artery of the descending colon via pressure sensor introduced in the artery and doppler
    3. Measurement of saturation via a saturation sensor
    4. Measurement of systemic blood pressure using a tension cuff
  * Time 2: after inferior mesenteric artery release restoring arterial blood flow in the artery and at least 10min since ICG injection of time 1 to obtain its clearance. same parameters mesured
  Interventions: Procedure: Clamping and restauration of arterial blood of the inferior mesenteric artery

INTERVENTIONS:
Procedure: Clamping and restauration of arterial blood of the inferior mesenteric artery — * Injection of Indocynianine green (INFRACYANINE 25mg diluted in 10 mL solvent, IV injection of 3ml at a concentration of 2.5 mg/mL or 7.5 mg), (excluding NaCl), purge 10ml NaCl,
  * Camera model (STORZ)
  * Camera/target distance: 5cm
  * Camera recording time (since Indocynianine green injection): 2 to 5 min with temporal identification of the injection time.
  Extracorporeal evaluation (by mini laparatomy extraction in colorectal surgery minimally invasive, by laparotomy in case of ovarian cancer with lights of the room switched off (laparotomy)

SUMMARY:
Colorectal cancers and ovarian cancers are respectively the 2nd and 5th cause of cancer mortality in France.

Surgical resection is a crucial step in the therapeutic management of colorectal cancers. For advanced ovarian cancers, the objective of cytoreductive surgery is to obtain complete macroscopic resection with no visible residual disease. One or more digestive resections are often required to achieve this goal of complete surgery (usually a modified posterior pelvic exenteration with colorectal resection).

A ligation of the inferior mesenteric artery at its origin is classically performed in left colectomies and rectal resection for colorectal cancers. This allows the resection of the colorectal segment with a complete mesocolic lymphadenectomy until the origin of the inferior mesenteric artery and a good mobilization of the descending colon to allow its anastomosis to the underlying rectal stump. This ligation of the inferior mesenteric artery at its origin is also frequently performed in cases of modified posterior pelvic exenteration for ovarian cancer.

Recently, several studies suggest that arterial ligation of the inferior mesenteric artery could be performed below the emergence of the left colic artery. Its preservation requiring a meticulous vascular dissection would allow a better vascularization of the descending colon and of the colorectal anastomosis without affecting the carcinologic quality of the resection and the number of resected lymph-nodes. Indeed, the most feared complication during colorectal anastomosis is the anastomotic leakage whose rates are on average 15% in rectal cancer with low anastomosis and 6% in ovarian cancers.

Verifying the adequate vascularization of the descending colon before performing the colorectal anastomosis is a crucial step in reducing the risk of postoperative fistula. However, quantifying this vascularization is challenging, and several techniques can be used to assess it. The gold standard technique involves measuring arterial pressure using a catheter inserted into the marginal artery of the descending colon. Other non-invasive techniques also use Doppler studies to calculate pressure in the marginal artery or assess oxygen saturation using a sterile sensor.

Studies have shown that the use of indocyanine green in colorectal surgery, particularly to evaluate perfusion before the creation of an anastomosis, significantly reduces the rate of anastomotic leakage. Indocyanine green is a fluorescent dye that, after intravenous injection, binds to plasma proteins and allows tissue perfusion to be visualized using a fluorescence system.

The objective of this project is to show that the preservation of the left colic artery is possible and allows a better vascularization of the descending colon before colorectal anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Male/ female aged over 18 years,
* Histologically proven left colon or rectal adenocarcinoma OR ovarian carcinoma (with potential colorectal resection),
* Scheduled surgery for left colic or rectal carcinoma// Scheduled surgery for ovarian carcinoma with potential colorectal resection,
* Surgical indication of colo-rectal resection validated in RCP and confirmed during the operative exploration (ovarian cancer,
* WHO Status < 3
* Patient who has given informed, written and express consent,
* Patient (s) affiliated to a French social security.

Exclusion Criteria:

* Contraindication to indocyanine green: thyroid adenoma, hyperthyroidism, hypersensitivity or allergy to one of the components, severe renal failure (GFR <30 ml/min/1.73m2),
* Patient with a history of abdominal vascular surgery
* Patient (e) not having left colic artery on vascular mapping of preoperative abdominal-pelvic scanners,
* Patient whose regular follow-up is not possible for psychological, family, social or geographical reasons,
* Patient (s) under guardianship, curatorship or safeguard of justice,
* Pregnant and/or breastfeeding patient,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-27 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of the variation in vascularization of the descending colon with or without clamping of the inferior mesenteric artery quantified by the method selected during the exploratory phase of the primary endpoint. | During the surgery
  Measurement of vascularization at the end of the descending colon with and without clamping the inferior mesenteric artery at its origin (interrupting arterial flow in the left colic artery) according to the quantification method selected in the exploratory evaluation phase.
  * If Indocyanine green intraveinous injection: measurement of decrease in staining time and increase in intensity
  * If Blood Pressure by catheter, doppler or saturation: percentage increase all the measures will define the same measure, that is to say, the vascularization of the descending colon

SECONDARY OUTCOMES:
Quantification of blood pressure in the marginal artery of the colon descending after clamping of the IMA at its origin then without clamping of the left colic artery by the other three method | During the surgery
  Measurement of blood pressure after catheterization of the marginal artery of the descending colon. Measurement of systemic blood pressure at the same time. The measurement will be performed using an arterial catheter.
Study of the anatomy of the lower mesenteric artery and its branches after arterial reconstruction of scanner performed preoperatively. | Before the surgery. At the baseline
  On the intraoperative Thoraco Abdomino Pelvis scanner, measure of the diameter in mm of the left colic artery.
Study of the anatomy of the lower mesenteric artery and its branches after arterial reconstruction of scanner performed preoperatively. | Before the surgery. At the baseline
  On the intraoperative Thoraco Abdomino Pelvis scanner, measure the distance in mm between the origin of the inferior mesenteric artery.
Study of the anatomy of the lower mesenteric artery and its branches after arterial reconstruction of scanner performed preoperatively. | Before the surgery. At the baseline
  On the intraoperative Thoraco Abdomino Pelvis scanner, evaluate the presence of dividing branches.
Evaluation of the operative parameters (operating time). | During the surgery
  operating time : in minutes: time between opening and closing of the skin
Evaluation of the operative parameters (duration of dissection of the inferior mesenteric artery). | During the surgery
  inferior mesenteric artery dissection time : in minutes: time between the beginning of the dissection of the I and completion
Evaluation of the operative parameters (duration of dissection of the left colic artery). | During the surgery
  left colic artery dissection time : in minutes:MA time between the beginning of the artery dissection and completion
Evaluation of the operative parameters (intraoperative bleeding). | During the surgery
  intraoperative bleeding in mL: estimated total volume of blood, measured by aspiration and impregnated compresses.
Evaluate postoperative parameters (within 30 days of surgery): rate of anastomotic leakage, rate of surgical recovery, duration of bowel function recovery. | 30 days after the surgery
  Data recovery within 30 days of surgery: anastomotic leakage rate (number of patients with anastomotic leakages confirmed by scan within 30 days of surgery), surgical recovery rate (number of patients for whom a re-intervention was necessary following a postoperative complication) and duration of bowel recovery (in days, defined by the 1st gas/stool emission after the intervention, defined by a clinical assessment of the surgeon).
Number of resected lymph-nodes. | 30 days after the surgery
  Total number of lymph nodes taken from the surgical specimen analysed in anatomopathology
Percentage of conservation of the colic artery. | 30 days after the surgery
  Success Percentage of conservation of the colic artery among included patient in the study.

OTHER OUTCOMES:
Determine the most appropriate measurement parameter to verify and quantify the vascularization of the descending colon among the following 4 methods | During the surgery for the 15 first patient
  * The measureof Blood pressure in the marginal artery of the colon with a pressure sensor introduced into the artery through a catheter.
  * Intraveinous ICG injection with the measure of duration between bolus and maximum opacification of the colon and semi-quantitative assessment of the intensity of the green. The measure will focus on the variation between the injection time and the maximum opacification (visual measurement) of the colon.
  * The measure of saturation in the marginal artery of the descending colon by a saturation sensor. The measure will be on the saturation variation in the artery.
  * The measure of BP in the marginal artery of the colon by Doppler. The measurement will be on the variation of pressure in the artery.
  This first phase will establish the best method to observe an increase in revascularization between clamped and non-clamped time
  all the measures will define the same measure, that is to say, the vascularization of the descending colon

CONTACTS AND LOCATIONS:
Locations (1):
- Icm Val D'Aurelle, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients All participant data collected during the trial, after coding by an inclusion number, 1st letter of the surname and first name can be shared.
  Participant data will be available upon request and with the completion of a contract between the sponsor and the applicant.
  The study protocol, the statistical analysis plan and the analytical code may also be subject to data sharing under a transfer contract (EU-MCR).

REFERENCES:
- [Background] Classe JM, Joly F, Lecuru F, Morice P, Pomel C, Selle F, You B. Prise en charge chirurgicale du cancer epithelial de l'ovaire - premiere ligne et premiere rechute: Surgical management of epithelial ovarian cancer - first line and first relapse. Bull Cancer. 2021 Dec;108(9S1):S13-S21. doi: 10.1016/S0007-4551(21)00583-X. PMID 34955158
- [Background] Fan YC, Ning FL, Zhang CD, Dai DQ. Preservation versus non-preservation of left colic artery in sigmoid and rectal cancer surgery: A meta-analysis. Int J Surg. 2018 Apr;52:269-277. doi: 10.1016/j.ijsu.2018.02.054. Epub 2018 Mar 1. PMID 29501795
- [Background] Liu FC, Song JN, Yang YC, Zhang ZT. Preservation of left colic artery in laparoscopic colorectal operation: The benefit challenge. World J Gastrointest Surg. 2023 May 27;15(5):825-833. doi: 10.4240/wjgs.v15.i5.825. PMID 37342851
- [Background] Qu R, Li F, Zhou X, Fu W. Is the preservation of the left colic artery an ideal choice for patients undergoing colorectal cancer surgery? A meta-analysis. Asian J Surg. 2021 Oct;44(10):1347-1348. doi: 10.1016/j.asjsur.2021.07.001. Epub 2021 Jul 21. No abstract available. PMID 34303593
- [Background] Guidolin K, Covelli A, Chesney TR, Draginov A, Chadi SA, Quereshy FA. Apical lymphadenectomy during low ligation of the IMA during rectosigmoid resection for cancer. Surg Open Sci. 2021 Jun 23;5:1-5. doi: 10.1016/j.sopen.2021.06.002. eCollection 2021 Jul. PMID 34337371
- [Background] Li B, Wang J, Yang S, Shen J, Li Q, Zhu Q, Cui W. Left colic artery diameter is an important factor affecting anastomotic blood supply in sigmoid colon cancer or rectal cancer surgery: a pilot study. World J Surg Oncol. 2022 Sep 27;20(1):313. doi: 10.1186/s12957-022-02774-0. PMID 36163068
- [Background] Sabbagh C, Maggiori L, Panis Y. Management of failed low colorectal and coloanal anastomosis. J Visc Surg. 2013 Jun;150(3):181-7. doi: 10.1016/j.jviscsurg.2013.03.016. Epub 2013 May 9. PMID 23665058
- [Background] Valenti G, Vitagliano A, Morotti M, Giorda G, Sopracordevole F, Sapia F, Lo Presti V, Chiofalo B, Forte S, Lo Presti L, Tozzi R. Risks factors for anastomotic leakage in advanced ovarian cancer: A systematic review and meta-analysis. Eur J Obstet Gynecol Reprod Biol. 2022 Feb;269:3-15. doi: 10.1016/j.ejogrb.2021.12.007. Epub 2021 Dec 13. PMID 34942555
- [Background] Peiretti M, Bristow RE, Zapardiel I, Gerardi M, Zanagnolo V, Biffi R, Landoni F, Bocciolone L, Aletti GD, Maggioni A. Rectosigmoid resection at the time of primary cytoreduction for advanced ovarian cancer. A multi-center analysis of surgical and oncological outcomes. Gynecol Oncol. 2012 Aug;126(2):220-3. doi: 10.1016/j.ygyno.2012.04.030. Epub 2012 Apr 30. PMID 22555105
- [Background] Clayton RD, Obermair A, Hammond IG, Leung YC, McCartney AJ. The Western Australian experience of the use of en bloc resection of ovarian cancer with concomitant rectosigmoid colectomy. Gynecol Oncol. 2002 Jan;84(1):53-7. doi: 10.1006/gyno.2001.6469. PMID 11748976
- [Background] Rutegard M, Rutegard J. Anastomotic leakage in rectal cancer surgery: The role of blood perfusion. World J Gastrointest Surg. 2015 Nov 27;7(11):289-92. doi: 10.4240/wjgs.v7.i11.289. PMID 26649151
- [Background] Li Z, Zhou Y, Tian G, Liu Y, Jiang Y, Li X, Song M. Meta-Analysis on the Efficacy of Indocyanine Green Fluorescence Angiography for Reduction of Anastomotic Leakage After Rectal Cancer Surgery. Am Surg. 2021 Dec;87(12):1910-1919. doi: 10.1177/0003134820982848. Epub 2020 Dec 30. PMID 33377797
- [Background] Zhang W, Che X. Effect of indocyanine green fluorescence angiography on preventing anastomotic leakage after colorectal surgery: a meta-analysis. Surg Today. 2021 Sep;51(9):1415-1428. doi: 10.1007/s00595-020-02195-0. Epub 2021 Jan 11. PMID 33428000
- [Background] Pang HY, Chen XL, Song XH, Galiullin D, Zhao LY, Liu K, Zhang WH, Yang K, Chen XZ, Hu JK. Indocyanine green fluorescence angiography prevents anastomotic leakage in rectal cancer surgery: a systematic review and meta-analysis. Langenbecks Arch Surg. 2021 Mar;406(2):261-271. doi: 10.1007/s00423-020-02077-6. Epub 2021 Jan 7. PMID 33409585
- [Background] Landsman ML, Kwant G, Mook GA, Zijlstra WG. Light-absorbing properties, stability, and spectral stabilization of indocyanine green. J Appl Physiol. 1976 Apr;40(4):575-83. doi: 10.1152/jappl.1976.40.4.575. PMID 776922
- [Background] Ahn HM, Son GM, Lee IY, Park SH, Kim NS, Baek KR. Optimization of indocyanine green angiography for colon perfusion during laparoscopic colorectal surgery. Colorectal Dis. 2021 Jul;23(7):1848-1859. doi: 10.1111/codi.15684. Epub 2021 May 11. PMID 33894016
- [Background] Van den Hoven P, S Weller F, Van De Bent M, Goncalves LN, Ruig M, D Van Den Berg S, Ooms S, Mieog J, Ea Van De Bogt K, Van Schaik J, Schepers A, Vahrmeijer AL, Hamming JF, Van Der Vorst JR. Near-infrared fluorescence imaging with indocyanine green for quantification of changes in tissue perfusion following revascularization. Vascular. 2022 Oct;30(5):867-873. doi: 10.1177/17085381211032826. Epub 2021 Jul 28. PMID 34320878
- [Background] Son GM, Kwon MS, Kim Y, Kim J, Kim SH, Lee JW. Quantitative analysis of colon perfusion pattern using indocyanine green (ICG) angiography in laparoscopic colorectal surgery. Surg Endosc. 2019 May;33(5):1640-1649. doi: 10.1007/s00464-018-6439-y. Epub 2018 Sep 10. PMID 30203201
- [Background] Faber RA, Tange FP, Galema HA, Zwaan TC, Holman FA, Peeters KCMJ, Tanis PJ, Verhoef C, Burggraaf J, Mieog JSD, Hutteman M, Keereweer S, Vahrmeijer AL, van der Vorst JR, Hilling DE. Quantification of indocyanine green near-infrared fluorescence bowel perfusion assessment in colorectal surgery. Surg Endosc. 2023 Sep;37(9):6824-6833. doi: 10.1007/s00464-023-10140-8. Epub 2023 Jun 7. PMID 37286750
- [Background] Pollmann L, Juratli M, Roushansarai N, Pascher A, Holzen JP. Quantification of Indocyanine Green Fluorescence Imaging in General, Visceral and Transplant Surgery. J Clin Med. 2023 May 18;12(10):3550. doi: 10.3390/jcm12103550. PMID 37240657
- See also: cancer environnement — https://www.cancer-environnement.fr/fiches/cancers/cancer-de-lovaire/
- See also: colorectal cancer — https://www.santepubliquefrance.fr/presse/2018/cancer-colorectal-18-000-deces-par-an
- See also: Related Info — https://www.snfge.org/tncd